CLINICAL TRIAL: NCT01349192
Title: Early MRSA Therapy in CF - Culture Based vs. Observant Therapy (Treat or Observe) (Star-TOO - STaph Aureus Resistance - Treat or Observe)
Brief Title: Early Methicillin-resistant Staphylococcus Aureus (MRSA) Therapy in Cystic Fibrosis (CF)
Acronym: STAR-Too
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim review showed a statistically significant treatment effect and the DMC recommended that the study be stopped with ongoing follow-up of enrolled subjects
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: CF Therapeutics Development Network Coordinating Center (Network); Seattle Children's Hospital (Other); Washington University School of Medicine (Other); University of Washington (Other); University of Colorado, Denver (Other); Baylor College of Medicine (Other); University of Alabama at Birmingham (Other); Cook Children's Medical Center (Other); University of Michigan (Other); University of Florida (Other); University of Texas Southwestern Medical Center (Other); Children's Hospital Medical Center, Cincinnati (Other); St. Louis Children's Hospital (Other)
Responsible Party: Principal Investigator, Marianne Muhlebach, MD, Professor, Pediatric Pulmonolgy, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STAR-too-10K0
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Cystic Fibrosis; Methicillin-resistant Staphylococcus Aureus
Keywords: MRSA; Cystic Fibrosis; Early Infection; Treatment
MeSH Terms: conditions — Cystic Fibrosis; Infections | interventions — Rifampin; Trimethoprim, Sulfamethoxazole Drug Combination; Minocycline; Mupirocin

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Although this is an open-label study, the PIs and operational study team will remain blinded to the study arm assignments of the aggregate study population and will not view aggregate study results by study arm until after database lock.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Subjects are treated with two oral antibiotics, topical antibiotics, and are instructed to use environmental decontamination techniques.
  Interventions: Drug: Rifampin; Drug: Trimethoprim/Sulfamethoxazole; Drug: Minocycline; Drug: Mupirocin; Drug: chlorhexidine gluconate oral rinse; Drug: 2% Chlorhexidine solution wipes; Behavioral: Environmental Decontamination
- Observational (No Intervention): Subjects are tracked and not treated for their MRSA. If the subject reaches a protocol defined exacerbation within the first 28 days then they will be treated per choice of their primary Pulmonologist.

INTERVENTIONS:
Drug: Rifampin — Adult Dose: 300mg twice daily for 14 days. Pediatric Dose: <40kg : 15mg/kg daily for 14 days divided every 12 hours.
  Other Names: Rifadin, Rimactane
  Arms: Treatment
Drug: Trimethoprim/Sulfamethoxazole — Adult Dose: 320/1600 orally twice daily for 14 days. Pediatric Dose: <40 kg : 8mg/kg trimethoprim / 40 mg/kg sulfamethoxazole twice a day for 14 days.
  Other Names: Bactrim, Septra
  Arms: Treatment
Drug: Minocycline — only subjects greater or equal to 8 years of age, who are not able to tolerate TMP/SMX or whose screening MRSA is resistant to TMP/SMX should be prescribed minocycline.
  Adult dose: 100 mg orally twice daily for 14 days Pediatric dose: < 50 kg : 2mg/kg orally twice daily for 14 days not to exceed 200mg per day.
  Other Names: Cleeravue-M, Dynacin, Minocin, Myrac, Solodyn, Vectrin
  Arms: Treatment
Drug: Mupirocin — 1 gram 2% nasal ointment generously applied to each nostril using a cotton swab twice daily for 14 days.
  Other Names: Bactroban, Centany
  Arms: Treatment
Drug: chlorhexidine gluconate oral rinse — for subjects able to swish without swallowing. 0.12% chlorhexidine gluconate oral rinse twice daily for 14 days.
  Arms: Treatment
Drug: 2% Chlorhexidine solution wipes — whole body wash solution wipes once daily for first 5 days.
  Arms: Treatment
Behavioral: Environmental Decontamination — wipe down high touch surfaces and medical equipment with surface disinfecting wipes daily for the first 21 days.
  wash all linens and towels in hot water once weekly for three weeks.
  Other Names: Sani-Cloth Plus
  Arms: Treatment

SUMMARY:
Purpose: There has been a recent, rapid increase in prevalence of Methicillin-resistant Staphylococcus aureus (MRSA) among patients with Cystic Fibrosis (22% across US CF centers in 2009). Some epidemiologic studies suggest possible worse outcomes, a recent analyses showing this with chronic but not intermittent MRSA. Given the chronic difficult to treat lung infections in CF it is unclear how the onset of MRSA should be approached. This randomized, controlled, interventional study seeks to determine if an early eradication protocol is effective for eradication of MRSA and will provide an opportunity to obtain data regarding early clinical impact of new isolation of MRSA.

Participants: Cystic fibrosis patients with new isolation of MRSA from their respiratory culture on a routine clinic visit.

Procedures (methods): Randomized, open-label, multi-center study comparing use of an eradication protocol to an observational group who receives the current standard of care i.e. treatment for MRSA only with pulmonary exacerbations.

DETAILED DESCRIPTION:
The STAR-too study is a randomized, open label, multi-center study in CF patients with new MRSA isolated from the respiratory tract (sputum or oropharyngeal (OP) swab). The purpose of the study is to compare use of a two week eradication treatment protocol to an observational group treated for MRSA only when respiratory symptoms meet the criteria for a protocol defined pulmonary exacerbation during the first 28 days of the study. A total of 90 participants, four years of age or older, with new MRSA infection are planned to be randomized in a 1:1 fashion to either the treatment arm or to the observational control arm. Randomization is stratified by age, P. aeruginosa status at screening and site. Each participant randomized to the treatment arm receives two oral antibiotics for 14 days, topical antibacterial treatment of skin and nares, and a three week environmental decontamination for high risk areas and equipment. Each participant randomized to the observational control arm is followed clinically with usual care except to treat new or worsening pulmonary symptoms with antibiotics between screening and Day 28 only when participant meets criteria for a protocol defined exacerbation. Participants continue in the study for 6 months with study visits at Day 84 and Day 168 corresponding with their normal quarterly visits, this extension of observation provides additional data regarding natural history of MRSA infection and durability of the eradication protocol. The primary outcome is the proportion of participants with MRSA eradicated from respiratory tract cultures at Day 28. The secondary outcomes number of, and time to, pulmonary exacerbations, and use of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 4 and ≤ 45 years of age at the Screening Visit.
2. Documentation of a CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype and one or more of the following criteria:

   * sweat chloride ≥ 60 mEq/liter by quantitative pilocarpine iontophoresis test (QPIT)
   * two well-characterized mutations in the cystic fibrosis transmembrane conductive regulator (CFTR) gene
   * Abnormal nasal potential difference (change in NPD in response to a low chloride solution and isoproteronol of less than -5 mV)
3. First OR early repeat MRSA colonization defined as:

   * First MRSA colonization: first documented isolation of MRSA from respiratory tract occurred ≤ 6 months prior to screening
   * OR Early repeat MRSA colonization:

   MRSA was previously isolated from the respiratory tract (≤ 2 times), but this was followed by at least 1 year of documented negative cultures for MRSA as noted below:

   -- At least 2 cultures performed at least 3 months apart to document 1 year of culture negativity. Each of these cultures should be documented to have been collected at least 1 week after end of any antibiotic prescription with MRSA activity.

   Patient again recently positive for MRSA from the respiratory tract (within 6 months prior to screening)
4. Clinically stable with no significant changes in health status within the 14 days prior to screening
5. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study

A repeat culture from the respiratory tract is obtained at screening but does not have to be positive to be able to enter the study.

Exclusion Criteria:

1. Received antibiotics with activity against MRSA within 28 days prior to screening (see study manual for list of antibiotics)
2. Use of an investigational agent within 28 days prior to screening
3. For subjects ≥ 6 years of age: FEV1 at screening < 30% of predicted for age based on the Wang (males < 18 years, females < 16 years) or Hankinson (males ≥ 18 years, females ≥ 16 years) standardized equations
4. MRSA from the screening culture resistant to rifampin OR resistant to both TMP/SMX and minocycline
5. History of intolerance to oral rifampin, or topical chlorhexidine or mupirocin
6. History of intolerance to both TMP/SMX and minocycline
7. < 8 years of age and either allergic or intolerant to TMP/SMX or screening MRSA resistant to TMP/SMX
8. ≥ 8 years of age and allergic or intolerant to TMP/SMX and screening MRSA resistant to minocycline
9. ≥ 8 years of age and allergic or intolerant to minocycline and screening MRSA resistant to TMP/SMX
10. For females of child bearing potential: pregnant, breastfeeding, or unwilling to use barrier contraception through Day 15 of the study
11. Abnormal renal function at Screening, defined as estimated creatinine clearance <50 mL/min using the Cockcroft-Gault equation
12. Abnormal liver function at the time of screening, defined as ≥2x upper limit of normal (ULN), of serum aspartate transaminase (AST) or serum alanine transaminase (ALT)
13. History of solid organ or hematological transplantation
14. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Ages: 4 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne S Muhlebach, MD, Principal Investigator — UNC Children's Hospital; Chris Goss, MD, Principal Investigator — University of Washington
Locations (13):
- United States (13):
  - The Children's Hospital-University of Birmingham, Birmingham, Alabama
  - The Children's Hospital, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - University of Michigan Health System, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota Minneapolis, Minneapolis, Minnesota
  - St. Louis Children's Hospital, St Louis, Missouri
  - N.C Memorial Hospital and N.C Children's Hospital, Chapel Hill, North Carolina
  - CFF Care Center & Pediatric Program Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lo DK, Muhlebach MS, Smyth AR. Interventions for the eradication of meticillin-resistant Staphylococcus aureus (MRSA) in people with cystic fibrosis. Cochrane Database Syst Rev. 2022 Dec 13;12(12):CD009650. doi: 10.1002/14651858.CD009650.pub5. PMID 36511181
- [Derived] Muhlebach MS, Beckett V, Popowitch E, Miller MB, Baines A, Mayer-Hamblett N, Zemanick ET, Hoover WC, VanDalfsen JM, Campbell P, Goss CH; STAR-too study team. Microbiological efficacy of early MRSA treatment in cystic fibrosis in a randomised controlled trial. Thorax. 2017 Apr;72(4):318-326. doi: 10.1136/thoraxjnl-2016-208949. Epub 2016 Nov 15. PMID 27852955

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted from April 1, 2011 to September 2014 at 14 CF Foundation accredited care centers in the United States.
Groups:
- Treatment: Oral antibiotics:
  1. Rifampin: Adult Dose: 300mg twice daily for 14 days. Pediatric Dose: <40kg : 15mg/kg daily for 14 days divided every 12 hours.
  2. Trimethoprim/Sulfamethoxazole: Adult Dose: 320/1600 orally twice daily for 14 days.
  Pediatric Dose: <40 kg : 8mg/kg trimethoprim / 40 mg/kg sulfamethoxazole twice a day for 14 days.
  Alternative 2) Minocycline: subjects greater or equal to 8 years unable to take TMP/SMX or whose screening MRSA is resistant to TMP/SMX are prescribed minocycline.
  Adult dose: 100 mg orally twice daily for 14 days Pediatric dose: < 50 kg : 2mg/kg orally twice daily for 14 days max 200mg per day.
  Topical:
  Mupirocin: 1 gram 2% nasal ointment twice daily for 14 days.
  Topical: 0.12% chlorhexidine gluconate oral rinse: for 14 days.
  Environmental disinfection of high use areas
Period: Overall Study
Arm/Group | Treatment | Observational
Started | 24 | 23
Evaluable for Primary Endpoint | 22 | 19
Withdrawals | 3 | 6
Completed | 21 | 17
Not Completed | 3 | 6
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 1 | 3
Not completed — Failure to adhere to Protocol | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Observational | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.3 (6.6) | 10.5 (5.5) | 11.5 (6.1)
Age, Customized [Count of Participants; unit: Participants]
  Age Category: >=4 and <12 years | 13 | 15 | 28
  Age Category: >=12 and <18 years | 6 | 5 | 11
  Age Category: >18 years | 5 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 14 | 11 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity Combined: Caucasian | 19 | 17 | 36
  Race/Ethnicity Combined: Hispanic | 3 | 2 | 5
  Race/Ethnicity Combined: African-American | 1 | 1 | 2
  Race/Ethnicity Combined: Other | 1 | 1 | 2
CF Genotype [Count of Participants; unit: Participants]
  Delta F508 Homozygous | 6 | 12 | 18
  Delta F508 Heterozygous | 14 | 7 | 21
  Other | 4 | 2 | 6
  Unidentified | 0 | 0 | 0
FEV1 Percent of Predicted [Mean (Standard Deviation); unit: percent] — Percent of predicted forced expiratory volume in one second, based on Wang and Hankinson reference equations. Population: Lung function was assessed for the subset of participants that were ≥ 6 years old and able to reliably perform spirometry.
  percent
    number analyzed (Participants) | 20 | 17 | 37
    (all) | 98.5 (21.6) | 101.2 (11.8) | 99.8 (17.6)
FEV1 Percent of Predicted Category [Count of Participants; unit: Participants] — Population: Lung function was assessed for the subset of participants that were ≥ 6 years old and able to reliably perform spirometry.
  Participants
    number analyzed (Participants) | 20 | 17 | 37
    >=30% to <=50% | 1 | 0 | 1
    >50% to <=75% | 1 | 0 | 1
    >75% to <=100% | 7 | 5 | 12
    >100% | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: MRSA Culture Status
Description: Proportion of subjects with a negative culture for MRSA at Day 28.
Time Frame: Day 28
Population: The analysis population is defined as all of the participants who were randomized to a study arm and were assessed for the primary microbiologic efficacy endpoint at both baseline and Day 28.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment: Oral antibiotics:
  Rifampin: Adult Dose: 300mg twice daily for 14 days. Pediatric Dose: <40kg : 15mg/kg daily for 14 days divided every 12 hours.
  Trimethoprim/Sulfamethoxazole: Adult Dose: 320/1600 orally twice daily for 14 days.
  Pediatric Dose: <40 kg : 8mg/kg trimethoprim / 40 mg/kg sulfamethoxazole twice a day for 14 days.
  Alternative 2) Minocycline: subjects greater or equal to 8 years unable to take TMP/SMX or whose screening MRSA is resistant to TMP/SMX are prescribed minocycline.
  Adult dose: 100 mg orally twice daily for 14 days Pediatric dose: < 50 kg : 2mg/kg orally twice daily for 14 days max 200mg per day.
  Topical:
  Mupirocin: 1 gram 2% nasal ointment twice daily for 14 days. Topical: 0.12% chlorhexidine gluconate oral rinse: for 14 days. Environmental disinfection of high use areas
- Observation: Subjects are tracked and not treated for their MRSA. If the subject reaches a protocol defined exacerbation within the first 28 days then they will be treated per choice of their primary Pulmonologist.
Arm/Group | Treatment | Observation
Number analyzed (Participants) | 22 | 19
Participants | 18 | 5
Statistical Analysis 1: Comparison: Treatment vs Observation; Test type: Superiority; p = 0.0005, Chi-squared — The a priori threshold for statistical significance was 0.05; Proportion Difference (Final Values) = 0.56, 95% CI 2-sided [0.25 to 0.74] — Proportion difference was calculated as proportion negative for MRSA in the treatment group minus the proportion negative for MRSA in the observation group. 95% CI calculated using the Newcombe-Wilson method without continuity correction
Statistical Analysis 2: Comparison: Treatment vs Observation; Test type: Superiority; p = 0.0004, Chi-squared — Test includes adjustment for two interim reviews of efficacy data. The a priori threshold for statistical significance was 0.05; Proportion Difference (Final Values) = 0.525, 95% CI 2-sided [0.23 to 0.80] — Proportion difference was calculated as proportion negative for MRSA in the treatment group minus the proportion negative for MRSA in the observation group

2. Secondary Outcome: Antibiotic Use (Proportion of Subjects)
Description: Proportion of subjects treated with oral, inhaled, and IV antibiotics over the 6 month study.
Time Frame: 6 months
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Observation
Number analyzed (Participants) | 24 | 21
Participants | 17 | 13
Statistical Analysis 1: Comparison: Treatment vs Observation; Test type: Superiority; p = 0.5463, Chi-squared — The a priori threshold for statistical significance was 0.05; Proportion Difference (Final Values) = 0.09, 95% CI 2-sided [-0.18 to 0.34] — Proportion difference was calculated as proportion using antibiotics in the treatment group minus the proportion using antibiotics in the observation group. 95% CI calculated using the Newcombe-Wilson method without continuity correction

3. Secondary Outcome: Antibiotic Use (Days of Use Per Subject)
Description: Days of use of oral, inhaled, and IV antibiotics over the 6 month study.
Time Frame: 6 months
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment | Observational
Number analyzed (Participants) | 24 | 21
days | 21.9 (23.7) | 31.3 (44.0)
Statistical Analysis 1: Comparison: Treatment vs Observational; Test type: Superiority; p = 0.3683, t-test, 2 sided — The a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = -9.42, 95% CI 2-sided [-30.3 to 11.47] — Mean difference was calculated as mean days of antibiotic use in the treatment group minus the mean days of antibiotic use in the observation group

4. Secondary Outcome: Pulmonary Exacerbations
Description: Proportion of subjects with a protocol-defined pulmonary exacerbation (PE) between baseline and day 28 who are treated with antibiotics active against MRSA.
Time Frame: 28 days
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Observation
Number analyzed (Participants) | 24 | 21
Participants | 2 | 6
Statistical Analysis 1: Comparison: Treatment vs Observation; Test type: Superiority; p = 0.1205, Chi-squared — The a priori threshold for statistical significance was 0.05; Proportion Difference (Final Values) = -0.20, 95% CI 2-sided [-0.42 to 0.03] — Difference was calculated as proportion with a PE treated with MRSA active antibiotics in the treatment group minus the analogous proportion in the observation group. 95% CI calculated using the Newcombe-Wilson method without continuity correction

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Treatment | Observation
Serious Adverse Events (participants affected / at risk) | 1/24 | 1/21
Other Adverse Events (participants affected / at risk) | 19/24 | 13/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=24) | Observation (N=21)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=24) | Observation (N=21)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (7) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (8) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 1 (3)
Weight decreased (Investigations) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 9 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was completed prior to reaching the pre-specified number of participants as the Data Safety Monitoring committee observed that efficacy had been reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No